CLINICAL TRIAL: NCT01594684
Title: Cotavance™ Paclitaxel-Coated Balloon Versus Uncoated Balloon Angioplasty for Treatment of In-stent Restenosis in SFA and Popliteal Arteries COPA CABANA Study
Brief Title: Cotavance™ Paclitaxel-Coated Balloon Versus Uncoated Balloon Angioplasty for Treatment of In-stent Restenosis in SFA and Popliteal Arteries
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. med. Gunnar Tepe (Other)
Collaborators: Zeller (Unknown); Duda (Unknown); Albrecht (Unknown); Reimer (Unknown); Brechtel (Unknown); Diehm (Unknown); Strausinsky (Unknown); Jahnke (Unknown); Huppert (Unknown); Amendt (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Gunnar Tepe, Head of the Deparment of Diagnostic and Interventional Radiology, Klinikum Rosenheim
Organization: Klinikum Rosenheim (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EK 11108
Record Dates: First submitted 2012-05-03; First posted 2012-05-09 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Catherization
Keywords: restenosis; stent; drug eltuing balloon; peripheral arterial disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- drug eluting balloon (Active Comparator): treatment with drug eltuing balloon
  Interventions: Device: balloon angiolplasty - drug coated balloon (Cotavance, Medrad Inc.); Device: drug coated balloon inflation (Cotavance, Medrad Inc.)
- uncoated balloon (Placebo Comparator): treatment with uncoated balloon
  Interventions: Device: uncoated balloon (e.g. Admiral, Medtronic)
- double drug eluting balloon (Active Comparator): if treatment fails 30 days or later
  Interventions: Device: balloon inflation, drug coated balloon (Cotavance, Medrad Inc.)

INTERVENTIONS:
Device: balloon angiolplasty - drug coated balloon (Cotavance, Medrad Inc.) — balloon inflation
  Arms: drug eluting balloon
Device: drug coated balloon inflation (Cotavance, Medrad Inc.) — Balloon inflation
  Arms: drug eluting balloon
Device: uncoated balloon (e.g. Admiral, Medtronic) — balloon inflation
  Arms: uncoated balloon
Device: balloon inflation, drug coated balloon (Cotavance, Medrad Inc.) — ballon inflation
  Arms: double drug eluting balloon

SUMMARY:
In stent restenosis in peripheral artery disease (superficial and popliteal artery) either treated with uncoated or paclitaxel coated balloons.

ELIGIBILITY:
Inclusion Criteria:

1. In-stent restenosis or re-occlusion at the target lesion due to an interventional treatment > 3 months prior to enrollment.
2. Has evidence of ≥ 70% stenosis or occlusion in the SFA and/or popliteal confirmed by angiography that is 3-27 cm long.
3. Reference vessel diameter of 3 to 7 mm (reference vessel diameter = normal vessel diameter 1 cm proximal of the index lesion)
4. Patients (men and women) with PAD disease category 2 to 5 according to Rutherford classification.
5. Patient is eligible for an operative vascular intervention in case of complications during the procedure.
6. Female patients of child bearing potential must have a negative pregnancy test 7 days at theprior to the time of intervention.
7. Fully informed and signed consent must be obtained from each patient.
8. Patients must be willing and able to continue study participation following study procedure in order to ensure completion of all procedures and observations required by protocol.
9. Patient has evidence of at least one run off vessel that does not also require treatment for significant (≥ 50% stenosis or occlusion) stenosis during the index procedure to the ankle/foot of the limb to be treated. Treatment of infrapopliteal lesions must be staged at least 30 days before or after the index procedure.
10. If restnosis occurs in both arms 30 days or later (re-re-sternosis)- treament with two drug eluting balloons at the same location (double dose)

Exclusion Criteria:

1. Patients with more than two lesions in the target vessel requiring treatment (if the distance between two lesions is less than 2 cm, the lesions should be counted as one lesion). The second lesion should also be treated with either coated or uncoated balloons (according to the randomization)
2. Guidewire cannot cross lesion and/or an intentional subintimal approach in the stented lesion is required.
3. Patients with stent fractures grade 2-4.
4. Inflow lesion (proximal to the study lesion) with flow limitation not being successfully treated prior to treatment of the study lesion.
5. Acute thrombosis of the study lesion requiring lysis or thrombectomy prior to the treatment of the study lesion.
6. Acutely occurring symptoms with a lyses or an operation as a therapeutic option within the last 6 weeks within the study limb.
7. Potential loss of leg due to critical or acute ischemia.
8. No patent distal run-off vessel.
9. Aneurysm in the blood vessel intended for intervention in this study.
10. Blood platelet count < 100.000/mm3 or >700.000/mm3, leukocyte count < 3.000/mm3.
11. Contra-indication to anticoagulation, or any anti-platelet agent (e.g. aspirin, heparin, clopidogrel, ticlopidine, abciximab), or paclitaxel.
12. Known intolerance or contra-indication (e.g. severe hepatic (with ALAT and/or ASAT > 3 times the normal reference range) or renal (creatinine > 1.1 mg/dl in women and >1.5 mg/dl in men) to contrast agents which cannot be adequately pre-treated, e.g. with adequate hydration.
13. Severe illnesses such as cancer, liver or renal diseases, myocardial insufficiency leading to protocol deviations and/or a reduced life expectancy of less than 2 years.
14. Manifest hyperthyreosis.
15. Latent hyperthyreosis without adequate therapy, e.g., previous blocking with Natriumperchlorat (Irenat®).
16. Significant gastrointestinal hemorrhage within the previous 6 months prior to study participation.
17. History of hemorrhagic diathesis or coagulopathy or rejection of blood transfusions.
18. Medical reason against double anti-platelet therapy in anti-coagulated patient, e.g., receiving coumadine.
19. Any severe medical condition that might interfere with the interpretation of the data or result in an unacceptable risk for the patient's participation in the study, according to the judgment of the clinical investigator.
20. Female patient who is pregnant or lactating.
21. Patient under 18 years of age.
22. Participation in another clinical study up to 30 days prior to study entry.
23. Previous participation in the same trialstudy (only one leg can be treated within the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Late Lumen Loss (LLL) | 6 +/-2 months
  • Late lumen loss (difference between the angiographic minimum lumen diameter (MLD) immediately and at 6 months post index procedure) evaluated by quantitative angiography. Analysis will be performed by an independent Angiographic Core Laboratory

SECONDARY OUTCOMES:
• Procedural success | after intervention
  • Procedural success defined as ≤ 30% residual stenosis following the procedure at the target lesion (after prolonged dilation and stenting, if necessary)
Target lesion revascularization (TLR) | 6, 12 and 24 months
  • Clinically-driven target lesion revascularization (TLR) at 6, 12 and 24 months. Target lesion revascularization is defined as any reintervention or artery bypass graft surgery involving the target lesion.
Target vessel revascularization (TVR) | 6, 12 and 24 months
  • Target vessel revascularization (TVR) at 6, 12 and 24 months
Binary restenosis rate | 6, 12 and 24 months
  • Binary restenosis rate at 6, 12 and 24 months.
  o Binary restenosis defined as > 50% diameter stenosis via angiography or PVR ≥ 2.4 via duplex ultrasound. In cases where results are available for both angiography and duplex ultrasound, angiographic results (if conducted within follow-up window) will be used to determine binary restenosis
Rutherford category | 6, 12 and 24 months
  Change of Rutherford category post index procedure and at 6, 12, and 24 months as compared to baseline
Ancle Brachial index (ABI) | 6, 12 and 24 months
  • Change in ABI at 6, 12, and 24 months as compared to baseline
Late lumen loss (LLL) | 24 months
  • LLL at 24 months
Minimum lumen diameter (MLD) | 12 and 24 months
  • MLD at 12 and 24 months
Hospitalization | 6, 12 and 24 months
  • Hospitalization (extra days due to complications of the index procedure) and hospitalization between the follow-up visits due to the index lesion and index leg
safety | 30days
  • Evaluation of 30 days freedom from procedure related death, unplanned amputation, and TLR.
resteosis pattern | 6 and 24 months
  • Characterization of restenosis patterns between the two therapies
Target lesion revascularization (TLR), clinical success and angiographic outcome (restenosis rate, late lumen loss) after second therapy | after intervention, 6, 12 and 24 months
  clinical success, restensosis, TLR and LLL after second use of drug eluting balloons if initial therapy failed 30 days or later

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Herzzentrum Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Tepe, Rosenheim, Baden-Wurttemberg
  - Uniklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Jüdisches Krankenhaus, Berlin, DE
  - Klinikum Neukölln, Berlin, DE
  - Klinikum Neumünster, Neumünster, Schleswig-Holstein

REFERENCES:
- [Derived] Tepe G, Schroeder H, Albrecht T, Reimer P, Diehm N, Baeriswyl JL, Brechtel K, Speck U, Zeller T. Paclitaxel-Coated Balloon vs Uncoated Balloon Angioplasty for Treatment of In-Stent Restenosis in the Superficial Femoral and Popliteal Arteries: The COPA CABANA Trial. J Endovasc Ther. 2020 Apr;27(2):276-286. doi: 10.1177/1526602820907917. Epub 2020 Feb 25. PMID 32096451